CLINICAL TRIAL: NCT01602198
Title: 24-week, Randomized, Double-blind, Placebo-controlled, Parallel Group Study of the Exelon® [Rivastigmine] Transdermal Patch in 120 APOE e4 Positive Amnestic MCI Patients
Brief Title: Study of Exelon Transdermal Patch in Amnestic Mild Cognitive Impairment Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study revised to use a different study medication and patient population.
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: AG022304
Record Dates: First submitted 2011-06-13; First posted 2012-05-18 (Estimated); Results first posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2016-12

CONDITIONS: Mild Cognitive Disorder; Mild Cognitive Impairment
MeSH Terms: conditions — Neurocognitive Disorders; Cognitive Dysfunction | interventions — Rivastigmine; Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exelon transdermal patch (Active Comparator): Exelon [rivastigmine] transdermal patch
  Interventions: Drug: Exelon [rivastigmine] transdermal patch
- Placebo transdermal patch (Placebo Comparator): Placebo transdermal patch
  Interventions: Drug: Placebo transdermal patch

INTERVENTIONS:
Drug: Exelon [rivastigmine] transdermal patch — Exelon patch 1/day for six months
  Other Names: Rivastigmine
  Arms: Exelon transdermal patch
Drug: Placebo transdermal patch — Placebo transdermal patch 1/day for 6 months
  Other Names: Placebo patch
  Arms: Placebo transdermal patch

SUMMARY:
The goal of this project is to determine if task-activated fMRI is sensitive to the central cholinergic deficit associated with Mild Cognitive Impairment.

DETAILED DESCRIPTION:
Clinical studies suggest that cholinesterase inhibitors (ChEIs) exert a cognitive benefit with chronic use among MCI and AD patients. Some studies also demonstrate a slight treatment benefit for persons who are APOE 4 positive. We propose to conduct a 24-week, randomized, double-blind, placebo-controlled, parallel group study of the Exelon® [rivastigmine] transdermal patch in 120 aMCI patients who have one or both APOE 4 alleles. Our preliminary analyses indicate that aMCI patients, even those who convert to AD, exhibit increased fMRI activation on our semantic memory activation task relative to not at-risk healthy participants and that increasing activation over time correlates with declines on neuropsychological testing. In addition, our preliminary data indicate that ChEI treated aMCI patients demonstrate normalization (i.e. reduction) in the magnitude of task-related neural activation over time relative to an untreated group. Furthermore, changes in fMRI magnitude demonstrated greater sensitivity to cholinergic modulation than changes on neuropsychological testing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of amnestic MCI
* In good general health with no diseases expected to interfere with the study
* Ability to undergo MRI
* Fluent in English
* Stable prescription dosages 1 month prior to testing
* Carrier of the APOE e4 allele (determined by blood draw at screening visit)

Exclusion Criteria:

* Neurological illness/conditions
* Medical illnesses/conditions that may affect brain function
* Prior history of use of any cholinesterase inhibitor
* Instable or severe cardiovascular disease or asthmatic condition

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Rao, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No data to share.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Transdermal Patch: Placebo transdermal patch
  Placebo patch: Placebo patch 1/day for 6 months
Period: Overall Study
Arm/Group | Exelon Transdermal Patch | Placebo Transdermal Patch
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exelon Transdermal Patch | Placebo Transdermal Patch | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 1 | 1
Gender [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in BOLD Response on Functional Magnetic Resonance Imaging (fMRI)
Time Frame: baseline and 6 months
Population: Trial was terminated prematurely after enrollment of only 1 participant. Sample size is insufficient for BOLD response analysis.
Arm/Group | Exelon Transdermal Patch | Placebo Transdermal Patch
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the study.
Arm/Group | Exelon Transdermal Patch | Placebo Transdermal Patch
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exelon Transdermal Patch (N=0) | Placebo Transdermal Patch (N=1)
High blood pressure (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No